CLINICAL TRIAL: NCT05369936
Title: Pain Perception: on Relationships Between Dental Anxiety and Olfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Ghada Khalifa, Professor of Maxillofacial Surgery and Diagnostic Science, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EA/3006/20018
Record Dates: First submitted 2021-12-20; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Dental Anxiety; Dental Pain; Essential Oil
Keywords: Dental Anxiety; Dental Pain; Emotional changes; Olfaction; Essential Oil; Lavender
MeSH Terms: conditions — Toothache; Anosmia | interventions — Aromatherapy; lavender oil

STUDY DESIGN:
Intervention Model Description: The patients will be divided into a control group in which the patients will be subjected to vapors of plain distal water, and lavender group where the patients will inhale vapors of the lavender oil to stimulate olfaction
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be performed according to patients' sequences where all odd numbers of patients will be incorporated into control group, while even numbers will be included in lavender group. The patients will not be informed about the type of the essential oil. T This was achieved by inserting lavender vaporizers in all setting rooms and clinics. So that the patients will believe that there is no extraordinary maneuver in the clinics. Also, all the dentists who treated the patients and evaluators who will interview the patients and questionnaires, will not be informed of the type of the essential oil which will be used. The statistician who will analyze the questionnaires will be informed that the study's groups are named as group A or B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender group (Experimental): On the day of the lavender group, after filling the first phase questionnaire, 20 drops of the lavender oil will be added to the electrical aromatherapy vaporizer near the patient's chair at a distance of 20 cm in the waiting room. After 20 minutes, the second phase questionnaire will be given to the patient, and then the patient will be transformed to dental clinics in which the lavender vaporizer will be placed near the dental unit at a distance of 20 cm. The vaporizer will be also prepared by adding 20 drops of the lavender which will be added added every 20 minutes until the dental sitting will be finalized, and the third questionnaire will be answered. At home, the patients will be asked to pour 3 drops of the lavender on a pad and inhale it for 5 minutes from 10 cm distance every one hour until they attend on the next day to answer the fourth questionnaire.
  Interventions: Other: Aromatherapy
- Placebo group (Placebo Comparator): The plain distal water vapors will be used as placebo, the good ventilation of the waiting room and clinics will be performed to ensure that the lavender scent is completely removed from the environment. The patients will inhale the vapors of the plain distal water
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — Lavender will be inhaled through three phases
  Other Names: Lavender
  Arms: Lavender group
Other: Placebo — Vapors of the distal water will be inhaled through three phases
  Other Names: Plain distal water
  Arms: Placebo group

SUMMARY:
the objective of this study is to evaluate the ability of olfaction in obtaining positive emotional and behavioral responses toward dental anxiety and pain in patients undergoing different dental procedures.

DETAILED DESCRIPTION:
All patients who meet inclusion criteria of the study will be given a written consent and enrolled into a randomized double-blinded controlled study (investigator and patients are blinded about the study). Patients will be divided into lavender and control groups. Patients in lavender group will subjected 2 % lavender vapors. In control group, patients will inhale distal water vapors

ELIGIBILITY:
Inclusion Criteria:

1. Adult females over 18 years,
2. Attending morning sessions of clinics (9 am)
3. Liable for administration of local anesthesia, tooth preparation either for filling procedures or crown preparations, endodontic treatment, teeth extraction, or subgingival scaling

Exclusion Criteria:

1. Males
2. Females who had allergies, bronchial asthma, common cold, pulmonary diseases, migraine, or taking antidepressants, anxiolytic drugs, opioids, or other medications that affect our results

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pain perception and anxiety is affected by gender. More common and exaggerated in females more than males
Enrollment: 350 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Anxiety score | 20 minutes before exposure to vapors
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Anxiety score | 20 minutes After exposure to vapors
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Anxiety score | 24 hours After exposure to vapors
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety

SECONDARY OUTCOMES:
Pain Score | 20 minutes before exposure to vapors
  A person rates their pain on a scale of 0 to 10 Zero means "no pain,"
  1 to 3 means mild pin 4 to 6 means moderate pain 7 to 10 means severe pain
Pain Score | 20 minutes after exposure to vapors
  A person rates their pain on a scale of 0 to 10 Zero means "no pain,"
  1 to 3 means mild pin 4 to 6 means moderate pain 7 to 10 means severe pain
Pain Score | 24 hours after exposure to vapors
  A person rates their pain on a scale of 0 to 10 Zero means "no pain,"
  1 to 3 means mild pin 4 to 6 means moderate pain 7 to 10 means severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Sarah AM Alkanan, Resident, Principal Investigator — Qusaiba Hospital, Qassim, Saudi Arabia; Hadeel S Alhaweri, Resident, Principal Investigator — Aljarirr Alshamali primary health care center, Qassim, Saudi Arabia; Ghada A Khalifa, Professor, Study Director — College of Dentistry, Qassim University, Saudi Arabia; Shaimaa MS Ata, Lecturer, Study Chair — College of Dentistry, Qassim University, Saudi Arabia
Locations (1):
- Ghada Amin Khalifa, Buraidah, Buraydah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
According to our authority regulations. It is not accepted to share date with other researchers